CLINICAL TRIAL: NCT03424915
Title: Integrative Profiling of Primary Breast Cancer on the Basis of Divergent Exercise Exposure
Brief Title: Exercise, Fitness and Tumor Profiling in Breast Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18-058
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue from the mastectomy or lumpectomy specimen may be obtained, may either acquire a fresh frozen research tumor and adjacent normal tissue sample or formalin fixed paraffin embedded (FFPE) tissue for molecular profiling Blood and research stool sample (if possible)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regular exercisers and non-exercising groups who have been diagnosed with breast cancer: There is no treatment on this study, it is a onetime assessment. exercisers: ≥120 minutes of vigorous-intensity aerobic exercise;There is no treatment on this study, it is a onetime assessment. non-exercisers: ≤ 30 minutes of moderate-intensity exercise per week.
  Interventions: Behavioral: Harvard Health Professionals survey; Other: Blood draw; Other: CPET Procedures; Other: stool sample; Procedure: Research Tissue sampling
- Regular exercisers who are at high risk of developing breast cancer: ≥120 minutes of vigorous-intensity aerobic exercise;
  Interventions: Behavioral: Harvard Health Professionals survey; Procedure: Research Tissue sampling

INTERVENTIONS:
Behavioral: Harvard Health Professionals survey — Participants will be asked a series of questions (using a validated questionnaire) to assess self-reported exercise exposure over the past 12 months.
Other: Blood draw — Participant will provide a blood sample
  Groups: Regular exercisers and non-exercising groups who have been diagnosed with breast cancer
Other: CPET Procedures — CPET with 12-lead ECG
  Groups: Regular exercisers and non-exercising groups who have been diagnosed with breast cancer
Other: stool sample — Research stool sample (within ±1 week of surgery), if possible
  Groups: Regular exercisers and non-exercising groups who have been diagnosed with breast cancer
Procedure: Research Tissue sampling — Sample of the tumor and normal breast tissue may be taken from the tissue removed during breast cancer surgery if there is enough tissue left over for research testing.

SUMMARY:
This study is designed to find out how engaging in regular exercise (or not) alters the biology of breast tumors as well as the normal tissue (if available) surrounding the tumor. The investigators hope that findings from this initial study will guide the design of future studies to examine how changes in exercise alter breast tumor biology.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1: Breast Cancer Patients

* Ages 21-80 years
* Female
* Histologically confirmed ER receptor positive (>1% staining), HER2 negative (FISH ratio <1.8), untreated operable breast cancer
* Stage I to II disease
* Scheduled for surgical resection by any type of mastectomy or lumpectomy at MSK
* Tumor size ≥1cm by preoperative imaging or physical examination
* Categorization into self-reported exercise history exposure classifications as follows: (1) exercising: ≥120 minutes of vigorous-intensity exercise/wk for the past 12 months, and (2) sedentary (non-exercising): ≤ 30 minutes of moderate-intensity exercise/week for the past months using the Harvard Health Professionals survey.(34)
* Ability to read and understand English
* Willing and able to comply with requirements of the protocol

Cohort 2: High-Risk Patients

* Women at high-risk of breast cancer, as defined by one of the following:

  * Cytologically confirmed atypical hyperplasia
  * confirmed LCIS
  * Being a carrier for BRCA1 and/or BRCA2
  * Predicted lifetime risk of breast cancer >20% based on family history
  * Predicted 10-year risk of breast cancer of ≥2.31%
  * Predicted 5-year risk of breast cancer ≥1.67%
* Aged 21-80 years old
* If a female of child-bearing potential, must not be pregnant or planning to become pregnant during the study.

  * Women <50 years old of child-bearing potential must have a negative pregnancy test (urine HCG or serum) within 14 days of enrollment.

Exclusion Criteria:

Cohort 1:

* Received any form of neoadjuvant treatment
* Presence of any other concurrent, actively treated malignancy
* Presence of metastatic disease
* If performing a CPET, any of the following contraindications:

  * Acute myocardial infarction within 3-5 days of any planned study procedures;
  * Unstable angina
  * Uncontrolled arrhythmia causing symptoms or hemodynamic compromise
  * Recurrent syncope
  * Active endocarditis
  * Acute myocarditis or pericarditis
  * Symptomatic severe aortic stenosis
  * Uncontrolled heart failure
  * Acute pulmonary embolus or pulmonary infarction within 3 months of any planned study procedures
  * Thrombosis of lower extremities
  * Suspected dissecting aneurysm
  * Uncontrolled asthma
  * Pulmonary edema
  * Respiratory failure
  * Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis).
* Mental impairment leading to inability to cooperate
* If performing a CPET, room air desaturation at rest ≤ 85%
* Any other condition or intercurrent illness that, in the opinion of the investigator, makes the participant a poor candidate for the study.

Cohort 2:

* Use of any selective estrogen receptor modulator or aromatase inhibitor within 6 months of consent, including, but not limited to: tamoxifen, raloxifene, arzoxifene, acolbifene, anastrozole, exemestane, and letrozole.
* Enrollment on an interventional investigational study
* Bilateral breast implants
* History of any of the following:

  * Invasive breast cancer
  * DCIS
* Any current invasive cancer diagnosis
* Metastatic malignancy of any kind
* If performing a CPET, any of the following contraindications:

  * Acute myocardial infarction within 3-5 days of any planned study procedures;
  * Unstable angina
  * Uncontrolled arrhythmia causing symptoms or hemodynamic compromise
  * Recurrent syncope
  * Active endocarditis
  * Acute myocarditis or pericarditis
  * Symptomatic severe aortic stenosis
  * Uncontrolled heart failure
  * Acute pulmonary embolus or pulmonary infarction within 3 months of any planned study procedures
  * Thrombosis of lower extremities
  * Suspected dissecting aneurysm
  * Uncontrolled asthma
  * Pulmonary edema
  * Respiratory failure
  * Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis).
* Mental impairment leading to inability to cooperate
* If performing a CPET, room air desaturation at rest ≤ 85%
* Any other condition or intercurrent illness that, in the opinion of the investigator, makes the participant a poor candidate for the core biopsy or the study.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Study Population: MSK clinic
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
differences in DNA somatic mutational profile | 2 years
  Eight-μm-thick representative sections of the fresh-frozen sample will be microdissected with a needle under a stereomicroscope (Olympus SZ61), to ensure >70% of tumor cell content as previously described.(36) Matched germline DNA will be microdissected from adjacent normal breast tissue (if available) for each case; to avoid the possibility of morphologically appearing non-neoplastic cells harboring somatic mutations; we will prioritize the microdissection of stromal cells and avoid normal breast ducts and lobules.
differences in RNA sequencing | 2 years
  The initial analysis will focus on immune signatures (i.e., immune activation, as well as preexisting immune and related signatures) characterization using RNA-seq

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent and Follow-up), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and Follow-up), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Follow-up), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and Follow-up), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and Follow-up), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (Consent and Follow-up), New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Follow-up), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm